CLINICAL TRIAL: NCT05020210
Title: Effect of Early Treatment With Sivelestat Sodium on Lung Function and Inflammatory Response of ARDS Patients
Brief Title: Effect of Early Treatment With Sivelestat Sodium in ARDS Patients
Acronym: siv-ARDS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Guangdong No.2 Provincial People's Hospital (Other); Foshan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-187
Record Dates: First submitted 2021-07-27; First posted 2021-08-25 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-06

CONDITIONS: ARDS; Inflammatory Response
Keywords: sivelestat; ARDS; Inflammatory Response; lung function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sivelestat Sodium group: Patients treated with Sivelestat Sodium within 72 hours of the diagnosis of ARDS.
  Interventions: Drug: Sivelestat sodium
- Conventional treatment group: Patients not treated with Sivelestat Sodium/Normal Saline after the diagnosis of ARDS

INTERVENTIONS:
Drug: Sivelestat sodium — Patients were treated with Sivelestat Sodium within 72 hours of the diagnosis of ARDS.
  Groups: Sivelestat Sodium group

SUMMARY:
This study is a multicenter, prospective, observational cohort study. The subjects were patients who developed ARDS within the preceding 72h. They were divided into 2 groups based on the use of sivelestat sodium which was determined by the physician in charge based on the condition of the patients: sivelestat sodium group and conventional treatment group. 560 patients were planned to be enrolled, with 280 patients in each group. In the sivelestat sodium group, patients were treated with sivelestat sodium within 72h of the diagnosis of ARDS. After 5 days of sivelestat treatment, sivelestat treatment should be stopped if the oxygenation index is greater than 300mmHg for at least 3 consecutive times; otherwise, sivelestat treatment should be continued until the oxygenation index is greater than 300mmHg for at least 3 consecutive times; if sivelestat treatment is continued until the 14th day, the drug should be stopped regardless of the oxygenation situation. Baseline data and Murray lung injury score, inflammatory markers, routine test results, duration of ECMO use/length of hospital stay/length of ICU stay were recorded at 1, 3,5, and 7 days after patients were enrolled, and patients were followed up on the 28th and 90th days.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent;
* ≥18 years old;
* Patients developed ARDS in the preceding 72h;
* The total scores of the Murray lung injury scores were greater than 6 （When lung compliance was not measured, the total scores of the other three scores were greater than 4）;

Exclusion Criteria:

* Pregnancy or lactation;
* ARDS was diagnosed for more than 72 hours;
* Sivelestat sodium was used for treatment prior to enrollment;
* Patients with more than 3 extra-pulmonary organ injuries/failure;
* Severe chronic liver disease (Child-pugh grade C);
* Previous history of allergy to sivelestat sodium or any of its ingredients or preservatives;
* Patients whose primary disease cannot be effectively controlled;
* Patients judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients developed ARDS in the preceding 72h
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Murray lung injury score | change from admission to 7 days after enrollment
  The Lung Injury Score can be used to assess the adult patient for the extent of acute pulmonary damage. It can be used both at the onset of a lung disorder and during the course of the illness to monitor changing lung involvement.
  Parameters
  * chest X-ray evaluated for alveolar consolidation
  * ratio of the partial pressure of oxygen in arterial blood to the inspiratory fraction of oxygen
  * PEEP level if ventilated
  * respiratory compliance if known
The serum levels of IL-6 | change from admission to 7 days after enrollment

SECONDARY OUTCOMES:
Capillary leakage index | change from admission to 7 days after enrollment
  Ultrasound lung water score, capillary leakage index
Serum levels of leukocytes | change from admission to 7 days after enrollment
Serum electrolyte level | change from admission to 7 days after enrollment
renal function | change from admission to 7 days after enrollment
  The serum levels of creatinine
liver function | change from admission to 7 days after enrollment
  The serum levels of ALTand AST
myocardial injury indexes | change from admission to 7 days after enrollment
  The serum levels of cTnT, CK-MB
respiratory function | change from admission to 7 days after enrollment
  oxygenation index
infection and immunity | change from admission to 7 days after enrollment
  The serum levels of CRP
infection and immunity | change from admission to 7 days after enrollment
  The serum levels of PCT
infection and immunity | change from admission to 7 days after enrollment
  The serum levels of IL-10 and IL-1β
infection and immunity | change from admission to 7 days after enrollment
  The serum levels of TNF-α
coagulation function | change from admission to 7 days after enrollment
  The serum levels of APTT, PT, TT
coagulation function | change from admission to 7 days after enrollment
  The serum levels of INR
coagulation function | change from admission to 7 days after enrollment
  The serum levels of Fbg
Incidence of new organ insufficiency/failure after enrollment | up to 2 years
length of ventilation/length of hospital stay/length of ICU stay | up to 2 years
Mortality rate of in-hospital /28d/90d | 90 days after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Southern medical university Nanfang hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided